CLINICAL TRIAL: NCT04967170
Title: A Pilot, Randomized, Blinded, Controlled Study Evaluating Autologous Platelet-Rich Plasma for the Treatment of Vulvar Lichen Sclerosus
Brief Title: A Study to Evaluate Platelet Rich Plasma to Treat Vulvar Lichen Sclerosus
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jennifer R. Arthurs (Other)
Responsible Party: Sponsor-Investigator, Jennifer R. Arthurs, Sponsor-Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-009396
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Vulvar Lichen Sclerosus
MeSH Terms: conditions — Vulvar Lichen Sclerosus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet Rich Plasma Group (Experimental): Subject diagnosed with vulvar lichen sclerosus will receive Autologous Platelet-Rich Plasma (PRP)
  Interventions: Biological: Autologous Platelet-Rich Plasma (PRP)
- Sham Procedure Group (Sham Comparator): Subject diagnosed with vulvar lichen sclerosus will receive sham procedure of intralesional needle insertion without any injectate administered.
  Interventions: Other: Sham Procedure

INTERVENTIONS:
Biological: Autologous Platelet-Rich Plasma (PRP) — Two intralesional injections of approximately 5-6mL given approximately 6 weeks apart
  Arms: Platelet Rich Plasma Group
Other: Sham Procedure — Intralesional needle insertion without any injectate.
  Arms: Sham Procedure Group

SUMMARY:
The purposes of this study are to determine the safety and feasibility of autologous platelet-rich plasma for the treatment of vulvar lichen sclerosus, and to determine the efficacy of autologous platelet-rich plasma for the treatment of vulvar lichen sclerosus.

ELIGIBILITY:
Inclusion Criteria

* Female, ages 18 years and greater.
* Females of childbearing potential must have a negative pregnancy test prior to receiving the study drug and will agree to use adequate contraception (hormonal or barrier method or abstinence) from the time of screening to a period of 1 year following completion of the drug treatment cycle. Females of childbearing potential are defined as premenopausal and not surgically sterilized, or post-menopausal for fewer than 2 years. A urine pregnancy test will be performed prior to the administration of the study drug to confirm negative results. If the urine pregnancy test is positive, the study drug will not be administered and the result will be confirmed by a serum pregnancy test. Serum pregnancy tests will be performed at a central clinical laboratory, whereas urine pregnancy tests will be performed by qualified personnel using kit.
* Females becoming pregnant during the study will continue to be monitored for the duration of the study or completion of the pregnancy, whichever is longer. Monitoring will include perinatal and neonatal outcome. Any SAEs associated with pregnancy will be recorded.
* Diagnosis of Lichen Sclerosus.
* On a maintenance regimen of topical clobetasol for Lichen Sclerosus. Maintenance is defined as use of topical clobetasol 3 or fewer days per week. For patients with a new diagnosis of Lichen Sclerosus, they will complete 6 weeks of topical clobetasol ointment twice daily prior to enrollment in the study with transition to a maintenance regimen during study.
* Completed general physical evaluation with primary care provider within 12 months of enrollment.
* Full understanding of the requirements of the study and willingness to comply with protocol.
* Can provide written informed consent and complete HIPAA documentation after the nature of the study is fully explained and prior to any study-related procedure

Exclusion Criteria

* Pregnant or nursing, or planning on becoming pregnant during the study period.
* Clinically significant abnormal hematology (complete blood count with differential).
* Taking anticoagulant medications (e.g., warfarin, heparin) or clopidogrel (Plavix).
* Taking anti-rheumatic disease medication (including methotrexate or other antimetabolites) within 3 months prior to study enrollment.
* On chronic, immunosuppressive transplant therapy or having a chronic, immunosuppressive state, including use of systemic steroids/corticosteroids.
* Using topical steroids on affected area and unable to stop for the 6 week washout period prior to beginning the study. Topical steroid use will be exclusionary throughout week 12 of the study for patients randomized to receive PRP.
* Current tobacco product use, including nicotine patch or other nicotine products.
* Ongoing infectious disease, including but not limited to tuberculosis, HIV, hepatitis, and syphilis.
* Clinically significant cardiovascular (e.g., history of myocardial infarction, congestive heart failure or uncontrolled hypertension > 90 mmHg diastolic and/or 180 mmHg systolic), neurologic (e.g., stroke, TIA) renal, hepatic, or endocrine disease (e.g., diabetes).
* History of cancer/malignancy with the exception of adequately treated basal cell or squamous cell carcinoma of the skin within the last 5 years.
* History of blood dyscrasia, including but not limited to anemia, thrombocytopenia, and monoclonal gammopathy.
* Participation in a study of an experimental drug or medical device within 3 months of study enrollment.
* Known allergy to local anesthetics of other components of the study drug.
* History of or current evidence of alcohol or drug abuse or dependence, recreational use of illicit drug or prescription medications, or have use of medical marijuana within 30 days of study entry.
* Any illness or condition which, in the investigators' judgement will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 6 months
  Number of adverse events reported

SECONDARY OUTCOMES:
Change in patient-administered symptom score on Clinical Scoring System for Lichen Sclerosus | Baseline, 1 week, 6 weeks, 12 weeks, 3 months, 6 months
  Measured using the self-reported Clinical Scoring System for Lichen Sclerosus questionnaire that scores symptoms from 0 (no complaints) to 10 (extreme complaints)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Bodiford, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No